CLINICAL TRIAL: NCT06199310
Title: Feasibility of Using Resting Heart Rate and Step-counts From Patient-held Sensors During Clinical Assessment of Medical Emergencies (FUSE)
Brief Title: FUSE - Feasibility of Patient Held Sensors for Medical Emergencies
Acronym: FUSE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Betsi Cadwaladr University Health Board (Other Government)
Responsible Party: Principal Investigator, Dr Christian P Subbe, Consultant Physician, Senior Clinical Lecturer, Betsi Cadwaladr University Health Board
Other Study IDs: IRAS 321129
Record Dates: First submitted 2023-12-03; First posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: Medical Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators want to study how wearable devices can help track health changes in people when they are not feeling well. Normally, clinicians compare someone's vital signs, like heart rate, to average ranges from healthy folks. But what if clinicians compare these signs to the person's own normal when they were well? The investigators aim to check if wearable sensors can make this possible for many people. The investigators will look at heart rate differences when someone is admitted to the hospital compared to their stable days before. The investigators will see how their daily steps change a week before getting sick. This global study involves adults in emergency or acute care. Participation poses no risks, burdens, or immediate benefits to patients.

DETAILED DESCRIPTION:
Rationale:

Abnormalities of vital signs are quantified by comparison with 'usual' ranges, which are those observed in resting healthy populations. It might be more appropriate to compare vital sign values of an individual that is in distress with their own usual values recorded when they were stable and well. Wearable sensors might make this possible at scale.

Objectives:

* To quantify the difference between heart rate on admission to acute care compared to the previously recorded vital signs when 24 hours and 1 week prior of the same patient.
* The change in daily steps taken by the patient in the week prior to admission to acute care
* To assess the feasibility of using heart rate data from patients' own wearable sensors.

Study design:

An asynchronous, international, multicentre observational study using the Flash Mob Research design.

Study population:

Patients aged 18 years and up who present at the Emergency Department, Acute Medical Department or Ambulatory Emergency Care with an acute complaint.

Main study parameters/endpoints:

* The difference between heart rate measured on presentation to acute care services, and measured prior when stable and well.
* The daily number of steps taken in the week prior to presentation to acute care services.
* The proportion of patients assessed for an acute complaint who have recordings of vital signs measured before they became unwell.
* A description of the population that uses devices that collect vital signs in terms of sex, age-group, digital literacy, and their severity of illness on presentation (as measured by a standard set of vital signs and frailty).
* The devices used to measure vital signs before they became unwell, and the vital signs they measure.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

There is no burden or risk associated with participation to patients, and no immediate benefit.

ELIGIBILITY:
Inclusion Criteria:

A subject must meet all the following criteria:

* Have an acute presenting complaint
* Aged 18 years or older
* Uses any of the following: smart-watch, activity tracker, or other wearable monitoring device, a smart phone that collects data from other wearable device
* Ability to give informed consent

Exclusion Criteria:

* Unable to give informed consent, including patients with immediately life-threatening illness

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients presenting to hospital with a medical condition / complaint.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Hospital admission | Within 24 hours of assessment
  Proportion of patients admitted to hospital

SECONDARY OUTCOMES:
Change in heart rate | 1 week (+/- 1 day)
  Trends in heart rate (beats per minute) prior to admission to hospital
Change in step count | 1 week (+/- 1 day)
  Trends in step count (daily steps) in the week prior to admission to hospital

CONTACTS AND LOCATIONS:
Overall Officials: Christian Subbe, Principal Investigator — YSBYTY Gwynedd Hospital
Locations (1):
- Ysbyty Gwynedd, Bangor, United Kingdom